CLINICAL TRIAL: NCT07069712
Title: A Master Protocol of an Open-Label, Multi-Drug, Multi-Center, Phase II Platform Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Anti-tumor Activity of Novel Agents or Combinations as Perioperative Treatment in Participants With Locally Advanced Resectable Gastroesophageal Adenocarcinoma (GEMINI-PeriOp GC)
Brief Title: A Study of Novel Agents or Combinations as Perioperative Treatment in Participants With Locally Advanced Resectable Gastroesophageal Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D9804C00001; 2024-516909-23-00 (Other: EU CT Number)
Record Dates: First submitted 2025-06-24; First posted 2025-07-17 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Gastroesophageal Adenocarcinoma
Keywords: Locally Advanced Resectable Gastroesophageal Adenocarcinoma; Gastroesophageal Junction; Neoadjuvant Treatment; Perioperative Treatment; Gastric cancer; Immune checkpoint inhibitors; Chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — trastuzumab deruxtecan; Capecitabine; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Sub-study 1: AZD0901 plus Rilvegostomig and 5-FU or Capecitabine (Experimental): Participants will receive AZD0901 plus Rilvegostomig and 5-FU or Capecitabine as neoadjuvant combination therapy (pre-surgery period) and adjuvant combination therapy (post-surgery period) and later will receive Rilvegostomig as adjuvant monotherapy.
  Interventions: Drug: AZD0901; Drug: Rilvegostomig; Drug: Capecitabine; Drug: 5-Fluorouracil (5-FU)
- Sub-study 2: T-DXd plus Rilvegostomig and 5-FU or Capecitabine (Experimental): Participants will receive T-DXd plus Rilvegostomig and 5-FU or Capecitabine as neoadjuvant combination therapy (pre-surgery period) and adjuvant combination therapy (post-surgery period) and later will receive Rilvegostomig as adjuvant monotherapy.
  Interventions: Drug: Rilvegostomig; Drug: Trastuzumab Deruxtecan (T-DXd); Drug: Capecitabine; Drug: 5-Fluorouracil (5-FU)
- Sub-study 3: Rilvegostomig plus FLOT chemotherapy (Experimental): Participants will receive Rilvegostomig plus FLOT chemotherapy as neoadjuvant combination therapy (pre-surgery period) and adjuvant combination therapy (post-surgery period) and later will receive Rilvegostomig as adjuvant monotherapy.
  Interventions: Drug: Rilvegostomig; Drug: FLOT Chemotherapy

INTERVENTIONS:
Drug: AZD0901 — AZD0901 will be administered as an IV infusion.
  Other Names: Sonesitatug Vedotin
  Arms: Sub-study 1: AZD0901 plus Rilvegostomig and 5-FU or Capecitabine
Drug: Rilvegostomig — Rilvegostomig will be administered as an IV infusion.
  Other Names: AZD2936
Drug: Trastuzumab Deruxtecan (T-DXd) — T-DXd will be administered as an IV infusion.
  Other Names: DS-8201a
  Arms: Sub-study 2: T-DXd plus Rilvegostomig and 5-FU or Capecitabine
Drug: Capecitabine — Capecitabine (Fluoropyrimidine) will be administered orally as chemotherapy standard of care.
  Arms: Sub-study 1: AZD0901 plus Rilvegostomig and 5-FU or Capecitabine; Sub-study 2: T-DXd plus Rilvegostomig and 5-FU or Capecitabine
Drug: 5-Fluorouracil (5-FU) — 5-FU (Fluoropyrimidine) will be administered as an IV infusion as chemotherapy standard of care.
  Arms: Sub-study 1: AZD0901 plus Rilvegostomig and 5-FU or Capecitabine; Sub-study 2: T-DXd plus Rilvegostomig and 5-FU or Capecitabine
Drug: FLOT Chemotherapy — FLOT (5-FU, leucovorin, oxaliplatin, and docetaxel) Chemotherapy will be administered as an IV infusion.
  Arms: Sub-study 3: Rilvegostomig plus FLOT chemotherapy

SUMMARY:
GEMINI-PeriOp GC study will assess the safety, tolerability, pharmacokinetics (PK) and preliminary anti-tumor activity of novel agents or novel combinations as perioperative treatment in participants with locally advanced resectable gastric, gastroesophageal junction (GEJ), or esophageal adenocarcinoma who have not received previous treatment for the disease.

DETAILED DESCRIPTION:
This Phase II, open-label, multi-drug, multi-center platform study consists of individual sub-studies, each allows the assessment of multiple novel agents or novel combinations.

Participants will be assigned across 3 sub-studies, to have sufficient evaluable participants of the confirmed recommended dose by Safety Review Committee (SRC) for study intervention in each corresponding sub-study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented gastric, GEJ, or esophageal adenocarcinoma with resectable disease
* Participants who are CLDN18.2-positive and HER2-negative in Sub-study 1 or HER2-positive in Sub-study 2; no specific requirements for Sub-study 3
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ and bone marrow function
* Body weight > 35 kg

Exclusion Criteria:

* Participants had any prior anti-cancer treatment or surgery for the current gastric, GEJ, or esophageal cancer.
* Active or prior documented autoimmune or inflammatory disorders requiring systemic treatment with steroids or other immunosuppressive treatment
* Central nervous system (CNS) pathology
* Uncontrolled infections
* Participants with history of (non-infectious) interstitial lung disease (ILD)/pneumonitis, current ILD/pneumonitis, or suspected ILD/pneumonitis
* History of another primary malignancy
* Participants with any known or suspicious distant metastasis
* Uncontrolled hepatitis B and/or chronic or active hepatitis B
* Current or prior use of immunosuppressive medication within 14 days before the first dose of study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2027-01-28 (Estimated); Study Completion 2028-09-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Until sub-study completion, up to 38 months
  To assess the safety and tolerability of perioperative treatment.
Percentage of participants with pathological complete response (pCR) | Until sub-study completion, up to 38 months
  pCR is defined as no viable cancer cells, including lymph nodes after complete evaluation in the resected gastric, GEJ, or esophageal cancer specimen and all sampled regional lymph nodes following neoadjuvant treatment.

SECONDARY OUTCOMES:
Surgery completion rate as planned | Until sub-study completion, up to 38 months
  Surgery completion rate (including R0 and R1) as planned is defined as the percentage of participants who received intended gastrectomy or gastroesophagectomy as planned.
R0 resection (complete resection) rate as planned | Until sub-study completion, up to 38 months
  R0 resection (complete resection) rate as planned is the percentage of participants who received gastrectomy or gastroesophagectomy and had a confirmed margin-negative resection as planned.
Percentage of participants with tumor downstaging | Until sub-study completion, up to 38 months
  Tumor downstaging is defined as the lowering of the primary tumor (T) and/or regional lymph nodes (N) from pre-neoadjuvant clinical staging (pre-cTN) to post-neoadjuvant clinical staging (post-cTN) and to postoperative pathological staging (ypTN).
Event-free survival (EFS) | Until sub-study completion, up to 38 months
  EFS is defined as the time from the first dose of study intervention to documented Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) or non-RECIST 1.1 disease progression that precludes radical surgery or requires non-protocol therapy during the neoadjuvant through surgery period, or to documented RECIST 1.1 or biopsy-confirmed non-RECIST 1.1 recurrence or progression of disease during the adjuvant period, or death due to any cause at any time.
Disease-free survival (DFS) | Until sub-study completion, up to 38 months
  DFS is defined as the time elapsed from the date of the first post-surgery scan (ie, Adjuvant Baseline scan) until the date of first evidence of disease recurrence as determined by Investigator using RECIST 1.1 assessment (local or distant), or death due to any cause, whichever occurs first.
Objective response rate (ORR) | Until sub-study completion, up to 38 months
  ORR is defined as the percentage of participants who have a CR or PR as determined by Investigator using RECIST 1.1 at their latest assessment prior to surgery.
Overall survival (OS) | Until sub-study completion, up to 38 months
  OS is defined as the time from the first dose of the study intervention until the date of death due to any cause regardless of whether participant withdraws from treatment or receives another anti-cancer therapy.
Serum concentrations of study interventions | Until sub-study completion, up to 38 months
  To assess the serum concentrations of study interventions in participants receiving perioperative treatment.
Number of participants with positive anti-drug antibodies (ADA) | Until sub-study completion, up to 38 months
  To assess the immunogenicity of study interventions in participants receiving perioperative treatment.

CONTACTS AND LOCATIONS:
Locations (57):
- United States (6):
  - Research Site, Newark, Delaware
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Fairway, Kansas
  - Research Site, North Shores, Michigan
  - Research Site, New York, New York
  - Research Site, Pittsburgh, Pennsylvania
- Canada (2):
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- China (10):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changzhi
  - Research Site, Chengdu
  - Research Site, Fuzhou
  - Research Site, Hangzhou
  - Research Site, Kunming
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shijiazhuang
- Research Site, Tbilisi, Georgia
- Italy (7):
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Pisa
  - Research Site, Rozzano
  - Research Site, Udine
  - Research Site, Vicenza
- Japan (9):
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Hidaka-shi
  - Research Site, Kashiwa
  - Research Site, Kitaadachi-gun
  - Research Site, Kōtoku
  - Research Site, Nagoya
  - Research Site, Osaka
  - Research Site, Suita-shi
- Poland (2):
  - Research Site, Bialystok
  - Research Site, Warsaw
- Spain (8):
  - Research Site, Barcelona
  - Research Site, Elche
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Ourense
  - Research Site, Oviedo
  - Research Site, Santander
  - Research Site, Valencia
- Taiwan (4):
  - Research Site, Kaohsiung City
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Turkey (Türkiye) (4):
  - Research Site, Adapazarı
  - Research Site, Erzurum
  - Research Site, Fatih-Istanbul
  - Research Site, Istanbul
- United Kingdom (4):
  - Research Site, Bristol
  - Research Site, Dundee
  - Research Site, Headington
  - Research Site, Norwich

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/